CLINICAL TRIAL: NCT00328497
Title: A Phase 1-2 Safety and Efficacy Study of Panzem Nanocrystal Colloidal Dispersion Administered Orally in Combination With rhuMAb VEGF (Bevacizumab) in Patients With Locally Advanced or Metastatic Carcinoid Tumors
Brief Title: A Combination Study to Determine the Safety and Efficacy of Panzem NCD With Avastin in Metastatic Carcinoid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CASI Pharmaceuticals, Inc. (Industry)
Responsible Party: Carolyn F. Sidor, MD, MBA; Chief Medical Officer, EntreMed, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ME-CLN-002
Record Dates: First submitted 2006-05-18; First posted 2006-05-22 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Carcinoid Tumor
MeSH Terms: conditions — Carcinoid Tumor | interventions — 2-Methoxyestradiol; Bevacizumab

ARMS (1):
- 1 (Experimental): Panzem NCD will be dosed orally at a level of 1,000 mg, four times daily for 28 consecutive days and bevacizumab will be administered at a dose of 5 mg/kg as an intravenous bolus on Day 1 and Day 15 of the Treatment Period
  Interventions: Drug: Panzem (2-methoxyestradiol) NCD, Avastin (Bevacizumab)

INTERVENTIONS:
Drug: Panzem (2-methoxyestradiol) NCD, Avastin (Bevacizumab) — Panzem NCD 1,000 mg, four times daily for 28 consecutive days bevacizumab 5 mg/kg intravenous bolus on Day 1 and Day 15

SUMMARY:
This single center, open-label study will evaluate the safety and efficacy of Panzem (2-methoxyestradiol, 2ME2) Nanocrystal Dispersion (NCD) administered orally with recombinant human monoclonal antibody against vascular endothelial growth factor (bevacizumab) administered intravenously, in patients with locally advanced or metastatic carcinoid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented locally unresectable or metastatic carcinoid neuroendocrine tumor
* Measurable disease, according to RECIST, with at least one lesion that is unidimensionally measurable by conventional techniques to be greater than or equal to 2 cm in diameter, or by spiral CT to be greater than or equal to 1 cm in diameter
* 18 years or older

Laboratory data to include (next 7 bullet points):

* Aspartate aminotransferase(AST)and alanine aminotransferase (ALT)less than 2.5 times the upper limit of normal (less than 5 times upper limit of normal if liver metastasis present)
* Total bilirubin less than or equal to 2 mg/dL
* Serum creatinine less than or equal to 1.5 mg/dL
* Total white blood cell count greater than 3,500/mm3
* Absolute neutrophil count greater than or equal to 1,500/mm3
* International normalized ratio less then or equal to 1.5
* Platelets greater than or equal to 100,000/mm3
* Agree to use effective contraceptive methods
* Have an ECOG performance status of less than 2
* Life expectancy of greater than 12 weeks
* Ability to understand the requirements of the study, have provided written consent, and agree to abibe by the study restrictions

Exclusion Criteria:

* Pregnant or nursing, or refusal to use appropriate birth control
* An active infection
* Have a history of myocardial infarction or angina pectoris/angina equivalent in the last 12 months (the patient may be on antianginal medications if the symptoms can be fully controlled), or have uncontrolled congestive heart failure
* Have apparent central nervous system metastasis or carcinomatous meningitis
* Have had any active cancer in addition to the carcinoid tumor within the last 5 years, with the exception of superficial skin cancer
* Be receiving concurrent treatment with therapeutic doses of any anticoagulant including all forms of heparin and Coumadin
* Have current or a history of severe bleeding
* Uncontrolled / severe hypertension
* Previous history of nephrotic syndrome
* Urine protein: creatinine ratio greater than or equal to 1.0 at screening
* Have received radiotherapy or chemotherapy within the previous 4 weeks
* Participated in any clinical trial involving conventional or investigational drugs or devices within the previous 4 weeks
* Have had major surgery within 4 weeks or plan to undergo elective surgery during treatment
* Additional uncontrolled serious medical condition or psychiatric illness
* Have any condition that is likely to interfere with regular follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-05; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To assess the safety of Panzem NCD administered orally in combination with intravenous infusion of bevacizumab by evaluation of the frequency and severity of treatment emergent adverse events | Approximately monthly
To evaluate the objective tumor response rate by radiographic means using Response Evaluation Criteria in Solid Tumors | Approximately every 8 weeks
To determine the overall survival of patients with locally advanced or metastatic carcinoid tumors administered oral Panzem NCD in combination with intravenous infusion of bevacizumab | Approximately every 3 months

SECONDARY OUTCOMES:
To determine the progression-free survival of patients with locally advanced or metastatic carcinoid tumors administered oral Panzem NCD in combination with intravenous infusion of bevacizumab | Approximately every 3 months
To monitor the steady-state trough plasma levels of 2ME2 following 28-day dosing cycles of Panzem NCD when administered orally in combination with intravenous infusion of bevacizumab | Approximately monthly

CONTACTS AND LOCATIONS:
Overall Officials: Matthew H. Kulke, M.D., Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States